CLINICAL TRIAL: NCT04040933
Title: A 28-Day, Single-Center, Randomized, Comparator-Controlled, Proof-of-Principle Study to Assess Wound Healing Efficacies of Different Adhesive Bandages
Brief Title: A Study to Assess Wound Healing Efficacies of Different Adhesive Bandages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCSTOH001689; CCSTOH001689 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (8):
- Marketed Adhesive Bandage #1 (Active Comparator): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Marketed Adhesive Bandage #1
- Marketed Adhesive Bandage #2 (Active Comparator): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed only on Days 3, 5, 7, 9, 11, 13, 15, and 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Marketed Bandage #2
- Non-marketed Adhesive Bandage #1 (Active Comparator): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Non-Marketed Bandage #1
- Non-marketed Adhesive Bandage #2 (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Non-Marketed Bandage #2
- Non-marketed Adhesive Bandage #3 (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Non-Marketed Adhesive Bandage #3
- Non-marketed Adhesive Bandage #4 (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Non-Marketed Adhesive Bandage #4
- Non-marketed Adhesive Bandage #5 (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, bandage will be applied. This adhesive bandage will be changed daily from Day 1 through Day 16 and all wound sites will be uncovered from Day 16 to Day 28 for assessments.
  Interventions: Device: Non-Marketed Adhesive Bandage #5
- No Treatment (Uncovered, Negative Control) (No Intervention): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, no treatment will be applied as the wound will be kept uncovered as negative control.

INTERVENTIONS:
Device: Marketed Adhesive Bandage #1 — On the randomized wound site, a marketed adhesive bandage will be applied.
  Arms: Marketed Adhesive Bandage #1
Device: Marketed Bandage #2 — On the randomized wound site, a marketed adhesive bandage will be applied.
  Arms: Marketed Adhesive Bandage #2
Device: Non-Marketed Bandage #1 — On the randomized wound site, a non-marketed adhesive bandage will be applied.
  Arms: Non-marketed Adhesive Bandage #1
Device: Non-Marketed Bandage #2 — On the randomized wound site, a non-marketed adhesive bandage will be applied.
  Arms: Non-marketed Adhesive Bandage #2
Device: Non-Marketed Adhesive Bandage #3 — On the randomized wound site, a non-marketed adhesive bandage will be applied.
  Arms: Non-marketed Adhesive Bandage #3
Device: Non-Marketed Adhesive Bandage #4 — On the randomized wound site, a non-marketed adhesive bandage will be applied.
  Arms: Non-marketed Adhesive Bandage #4
Device: Non-Marketed Adhesive Bandage #5 — On the randomized wound site, a non-marketed adhesive bandage will be applied.
  Arms: Non-marketed Adhesive Bandage #5

SUMMARY:
The purpose of this study is to assess the wound healing efficacy (time to complete healing) of different adhesive bandages.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type II or III
* Uniform skin color on both volar forearms
* Generally in good health based on medical history reported by the participant
* -Individual has signed the Photographic Release and Informed Consent Documents along with (HIPAA) disclosure
* Willing to have temporary (semi-permanent) dot-tattoos applied to the volar forearms

Exclusion Criteria:

* Has known allergies, hypersensitivity, or adverse reactions to anesthetics, adhesive bandages, latex, wound treatment products, or any component/ingredient present in the Investigational Products (IPs)/auxiliary/ancillary products
* Has a known history of a blood-clotting disorder, keloid formation, or a cardiovascular, hepatic, or renal disease
* Presents with a skin condition that would, in the opinion of the PI or Study Physician, confound study results, increase risk to participant, or interfere with study evaluations
* Has excessive hair or tattoos on either volar forearm
* Has a known history of severe systemic immune system disorders
* Has self-reported Type 1 or Type 2 diabetes
* Has self-reported uncontrolled chronic diseases
* Is taking medication that would mask an adverse event, confound study results or alter/compromise the bleeding/healing process
* Is self-reported to be pregnant or planning to become pregnant
* Has a body mass index (BMI) above 35
* Is self-reported to be an alcohol or drug abuser
* Has participated in another clinical trial within 10 days
* Either is or lives with someone who is a current employee of any company that makes/markets adhesive bandages or first-aid products

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lily Jiang, PhD, Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (1):
- Thomas J. Stephens, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received all eight intervention at the same time on their forearms. At Screening (Visit 1; 3 to 7 days prior to Baseline), participants were provided with an auxiliary cleanser to use on their forearms and for all body cleansing in place of their regular body cleanser for the duration of the study. As planned, for all outcome measures, the results are reported for each bandage separately.
Groups:
- All Randomized Participants: All Participants with Fitzpatrick skin types II (burns easily; tans minimum)-III (burns moderately; tans gradually) with uniform skin color on forearms, minor wounds were created on forearms (four per arm) by a certified laser specialist received all eight intervention at the same time on the wounds created on forearms. Each wound site was subjected to one of eight randomly-assigned treatments included in an adhesive bandage that were: 1) a marketed adhesive bandage, 2) a marketed adhesive bandage (IP-benchmark control 1), 3) a non-marketed adhesive bandage (IP-benchmark control 2), 4-7) four non-marketed adhesive bandages (IP#1, IP#2, IP#3, IP#4), and 8) no treatment (uncovered, negative control). Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandages were not left on after a composite healing score of 8 was achieved.
Period: Overall Study
Arm/Group | All Randomized Participants
Started | 36
Treated | 36
Completed | 33
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Classification [Count of Participants; unit: Participants] — The Fitzpatrick skin classification is based on the skin's unprotected response to the first 30-45 minutes of sun exposure after a winter season without sun exposure. The classification is on a scale from I to VI where I = always burns easily; never tans and VI =Never burns; deeply pigmented.
  Participants
    Fitzpatrick Skin Classification - II | 24
    Fitzpatrick Skin Classification - III | 12

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Trans-Epidermal Water Loss (TEWL) Measurements
Description: Change from Baseline in TEWL was reported. TEWL is the passive transfer of water through stratum corneum and was measured for each wound site using Tewameter TM330T. TEWL is a non-invasive method to measure the integrity of stratum corneum barrier function. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. The probe was held in place on the skin for one measurement, for 40 sec, to ensure that a stable value has been established. The values of the last 10 sec are averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Day 0 (immediate after wound creation), Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14
Population: The Intent-to-Treat (ITT) set include all participants who received laser-induced wounds and started the study treatments. Here 'n' (number analyzed) included all evaluable participants analyzed at specified timepoints. As planned, for this outcome measure, the data was reported for each bandage separately.
Measure: Mean (Standard Deviation); unit: gram (g)/meter(m)^2/hour (g/m^2/hr)
Groups:
- Negative Control: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, no treatment was applied as the wound remained uncovered as negative control.
- Marketed Adhesive Bandage: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, marketed adhesive bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Marketed Adhesive Bandage IP-1 Benchmark Control 1: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, benchmark control 1 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Non-marketed Adhesive Bandage IP-Benchmark Control 2: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, benchmark control 2 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Non-marketed Adhesive Bandage IP #1: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, non-marketed IP#1 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Non-marketed Adhesive Bandage IP #2: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, non-marketed IP#2 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Non-marketed Adhesive Bandage IP #3: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, non-marketed IP#3 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
- Non-marketed Adhesive Bandage IP #4: Minor wounds were created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, non-marketed IP#4 bandage was applied. Bandages were changed daily/every other day until the wound reached a composite healing score of 8. The bandage was not left on after a composite healing score of 8 was achieved.
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
gram (g)/meter(m)^2/hour (g/m^2/hr)
  Day 0: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 0 | 39.27 (8.240) | 37.99 (10.050) |  | 39.57 (8.796) | 40.71 (9.284) | 39.06 (11.257) | 36.47 (8.789) | 38.74 (7.455)
  Day 1: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 1 | 39.70 (9.681) | 37.86 (11.667) |  | 36.30 (10.345) | 31.48 (11.157) | 34.96 (10.541) | 30.48 (8.864) | 40.14 (13.278)
  Day 2: number analyzed (Participants) | 35 | 35 | 0 | 35 | 35 | 35 | 35 | 35
  Day 2 | 25.31 (12.042) | 16.74 (11.902) |  | 14.08 (14.260) | 7.47 (6.792) | 11.68 (7.032) | 9.59 (6.051) | 19.55 (11.594)
  Day 3: number analyzed (Participants) | 35 | 35 | 33 | 35 | 35 | 35 | 35 | 35
  Day 3 | 12.80 (13.071) | 7.24 (9.361) | 2.33 (7.219) | 5.67 (11.081) | 4.60 (7.837) | 7.01 (5.896) | 5.37 (7.189) | 7.05 (8.513)
  Day 4: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 4 | 5.81 (10.096) | 2.65 (7.517) |  | 1.14 (9.210) | 5.09 (7.174) | 5.55 (11.303) | 3.71 (6.299) | 1.37 (7.505)
  Day 5: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 5 | 1.62 (7.636) | -0.21 (6.273) | -0.64 (6.867) | -1.47 (5.626) | 7.33 (8.932) | 4.56 (5.270) | 1.88 (5.856) | -2.42 (4.974)
  Day 6: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 6 | 5.40 (7.519) | 3.02 (7.410) |  | 3.73 (7.495) | 9.36 (7.163) | 6.56 (5.736) | 6.35 (5.221) | 1.04 (6.633)
  Day 7: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 33 | 33
  Day 7 | 1.89 (7.505) | 0.42 (6.266) | 4.33 (6.751) | 2.95 (14.523) | 9.45 (8.722) | 4.70 (5.079) | 3.51 (7.782) | -0.78 (6.177)
  Day 8: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 33 | 33 | 33
  Day 8 | 2.29 (6.629) | 2.22 (8.670) |  | 2.66 (7.315) | 9.24 (8.642) | 5.81 (5.742) | 5.16 (6.224) | 1.61 (8.170)
  Day 9: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 27 | 32
  Day 9 | 2.67 (8.623) | 3.60 (6.604) | 7.75 (7.210) | 3.15 (9.808) | 7.44 (6.151) | 6.50 (5.898) | 4.49 (6.350) | 1.60 (7.721)
  Day 10: number analyzed (Participants) | 33 | 33 | 0 | 33 | 32 | 32 | 28 | 32
  Day 10 | 0.61 (6.125) | 1.84 (7.714) |  | 0.81 (6.908) | 5.50 (6.187) | 3.79 (5.137) | 3.78 (6.538) | -0.48 (6.885)
  Day 11: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 11 | 1.30 (5.810) | 2.76 (7.082) | 4.20 (7.264) | 1.78 (7.190) | 5.60 (7.211) | 5.11 (4.491) | 6.89 (8.666) | 3.40 (13.542)
  Day 12: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 27 | 32
  Day 12 | 0.60 (7.181) | 0.47 (6.433) |  | 0.52 (5.468) | 1.21 (4.225) | 3.99 (6.655) | 3.66 (7.701) | 0.79 (8.074)
  Day 13: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 28 | 32
  Day 13 | 1.69 (6.367) | 1.96 (6.642) | 3.97 (7.060) | 0.59 (5.786) | 4.05 (5.576) | 5.68 (11.911) | 2.61 (6.831) | 1.13 (6.594)
  Day 14: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 27 | 32
  Day 14 | 0.91 (6.472) | 0.32 (5.469) |  | 0.55 (6.035) | 3.17 (4.744) | 4.33 (4.902) | 4.81 (12.362) | 1.97 (9.991)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline in TEWL measurements was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each baseline score within each treatment using paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p = 0.860, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.051, ANCOVA

2. Secondary Outcome: Change From Baseline in Clinical Grading of Wound Healing Parameter - Erythema
Description: Change from baseline in Clinical grading of wound healing parameter (erythema) was evaluated on a scale of 0 (no erythema) to 4 (severe erythema).
Time Frame: Day 0 (immediate after wound creation), Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Scores on a scale
  Day 0: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 0 | 1.04 (0.469) | 1.06 (0.459) |  | 1.08 (0.486) | 1.08 (0.486) | 1.07 (0.509) | 1.07 (0.550) | 1.06 (0.459)
  Day 1: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 1 | 3.03 (0.686) | 2.28 (0.760) |  | 2.07 (0.645) | 2.13 (0.740) | 2.10 (0.791) | 2.42 (0.849) | 2.03 (0.632)
  Day 2: number analyzed (Participants) | 35 | 35 | 0 | 35 | 35 | 35 | 35 | 35
  Day 2 | 3.51 (0.624) | 2.14 (0.703) |  | 1.83 (0.747) | 1.60 (0.746) | 1.79 (0.730) | 2.30 (0.769) | 1.81 (0.665)
  Day 3: number analyzed (Participants) | 35 | 35 | 33 | 35 | 35 | 35 | 35 | 35
  Day 3 | 3.50 (0.630) | 2.00 (0.795) | 1.62 (0.650) | 1.67 (0.696) | 1.29 (0.740) | 1.63 (0.668) | 2.40 (0.705) | 1.74 (0.657)
  Day 4: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 4 | 3.44 (0.600) | 1.82 (0.797) |  | 1.50 (0.728) | 1.03 (0.651) | 1.49 (0.702) | 2.25 (0.751) | 1.69 (0.718)
  Day 5: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 5 | 3.09 (0.691) | 1.72 (0.698) | 1.21 (0.687) | 1.51 (0.668) | 0.69 (0.508) | 1.53 (0.651) | 2.09 (0.633) | 1.76 (0.710)
  Day 6: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 6 | 2.82 (0.727) | 1.66 (0.648) |  | 1.31 (0.640) | 0.54 (0.528) | 1.28 (0.630) | 2.04 (0.829) | 1.62 (0.729)
  Day 7: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 7 | 2.41 (0.883) | 1.65 (0.764) | 0.79 (0.676) | 1.41 (0.645) | 0.56 (0.519) | 1.31 (0.779) | 1.94 (0.736) | 1.75 (0.846)
  Day 8: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 33 | 33 | 33
  Day 8 | 2.33 (0.747) | 1.45 (0.754) |  | 1.24 (0.675) | 0.62 (0.587) | 1.17 (0.633) | 1.68 (0.694) | 1.89 (0.726)
  Day 9: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 27 | 32
  Day 9 | 1.98 (0.805) | 1.38 (0.696) | 0.79 (0.685) | 0.98 (0.523) | 0.42 (0.378) | 0.95 (0.474) | 1.44 (0.560) | 1.67 (0.736)
  Day 10: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 27 | 32
  Day 10 | 1.88 (0.839) | 1.14 (0.628) |  | 0.88 (0.500) | 0.44 (0.390) | 0.86 (0.462) | 1.15 (0.569) | 1.52 (0.798)
  Day 11: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 11 | 1.67 (0.845) | 1.02 (0.492) | 0.56 (0.390) | 0.86 (0.472) | 0.39 (0.370) | 0.80 (0.455) | 1.13 (0.511) | 1.41 (0.798)
  Day 12: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 27 | 32
  Day 12 | 1.38 (0.650) | 0.88 (0.662) |  | 0.68 (0.411) | 0.32 (0.302) | 0.67 (0.433) | 0.91 (0.538) | 1.25 (0.660)
  Day 13: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 13 | 1.20 (0.624) | 0.70 (0.450) | 0.41 (0.384) | 0.61 (0.410) | 0.26 (0.309) | 0.58 (0.404) | 0.94 (0.543) | 1.16 (0.665)
  Day 14: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 28 | 32
  Day 14 | 1.23 (0.574) | 0.65 (0.537) |  | 0.53 (0.394) | 0.27 (0.333) | 0.42 (0.383) | 0.95 (0.567) | 1.05 (0.601)
  Day 15: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 15 | 1.09 (0.537) | 0.58 (0.417) | 0.30 (0.329) | 0.48 (0.385) | 0.17 (0.239) | 0.38 (0.311) | 0.72 (0.446) | 0.92 (0.555)
  Day 16: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 28 | 32
  Day 16 | 1.08 (0.486) | 0.56 (0.480) | 0.38 (0.331) | 0.47 (0.374) | 0.17 (0.239) | 0.36 (0.364) | 0.79 (0.535) | 0.86 (0.650)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline in Erythema measurements was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p = 0.259, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.451, ANCOVA

3. Secondary Outcome: Change From Baseline in Clinical Grading of Wound Healing Parameter - Edema
Description: Change from baseline in Clinical grading of wound healing parameter (edema) was evaluated on a scale of 0 (no edema) to 4 (severe edema).
Time Frame: Day 0 (immediate after wound creation), Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Scores on a scale
  Day 0: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 0 | 0.22 (0.326) | 0.21 (0.325) |  | 0.22 (0.347) | 0.22 (0.326) | 0.26 (0.439) | 0.28 (0.454) | 0.22 (0.347)
  Day 1: number analyzed (Participants) | 36 | 36 | 0 | 36 | 36 | 36 | 36 | 36
  Day 1 | 0.42 (0.439) | 0.01 (0.083) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 2: number analyzed (Participants) | 35 | 35 | 0 | 35 | 35 | 35 | 35 | 35
  Day 2 | 0.16 (0.291) | 0.00 (0.000) |  | 0.01 (0.085) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.085)
  Day 3: number analyzed (Participants) | 35 | 35 | 33 | 35 | 35 | 35 | 35 | 35
  Day 3 | 0.09 (0.191) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.085)
  Day 4: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 4 | 0.00 (0.000) | 0.00 (0.000) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 5: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 5 | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.171) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 6: number analyzed (Participants) | 34 | 34 | 0 | 34 | 34 | 34 | 34 | 34
  Day 6 | 0.00 (0.000) | 0.00 (0.000) |  | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.257) | 0.00 (0.000) | 0.00 (0.000)
  Day 7: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 7 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.171) | 0.00 (0.000) | 0.01 (0.086) | 0.00 (0.000) | 0.00 (0.000)
  Day 8: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 33 | 33 | 33
  Day 8 | 0.00 (0.000) | 0.00 (0.000) |  | 0.02 (0.087) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 9: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 27 | 32
  Day 9 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.087) | 0.00 (0.000) | 0.03 (0.174) | 0.00 (0.000) | 0.00 (0.000)
  Day 10: number analyzed (Participants) | 33 | 33 | 0 | 33 | 32 | 32 | 27 | 32
  Day 10 | 0.00 (0.000) | 0.00 (0.000) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 11: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 11 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 12: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 27 | 32
  Day 12 | 0.00 (0.000) | 0.00 (0.000) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.096) | 0.00 (0.000)
  Day 13: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 13 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.192) | 0.00 (0.000)
  Day 14: number analyzed (Participants) | 33 | 33 | 0 | 33 | 33 | 32 | 28 | 32
  Day 14 | 0.00 (0.000) | 0.02 (0.087) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.189) | 0.00 (0.000)
  Day 15: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 27 | 32
  Day 15 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 16: number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 32 | 28 | 32
  Day 16 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.094) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline in Edema measurements was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p > 0.999, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.739, ANCOVA

4. Secondary Outcome: Change From Baseline in Composite Scar Score
Description: Change from baseline in composite scar score was reported. It was calculated as the sum of the individual parameters on the Manchester Scar Scale (Color ranges 1 [perfect] to 4 [gross mismatch]), Finish ranges 1 [matte] to 2 [shiny], Contour ranges 1 [Flush with surrounding skin] to 4 [keloid], Distortion ranges 1 [none] to 4 [severe] and Texture ranges 1 [normal] to 4 [hard]). Composite Scar Scores range from 5 to 18, with 5 representing clinically best scars and 18 representing clinically worst scars.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 33 | 33
Scores on a scale | 2.09 (1.548) | 0.61 (0.496) | 0.33 (0.645) | 0.42 (0.502) | 0.24 (0.435) | 0.30 (0.467) | 0.88 (0.893) | 1.18 (1.103)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline in Composite Scar Score Measurements was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.053, ANCOVA

5. Secondary Outcome: Change From Baseline in Painful Score With Arm Resting by Side
Description: Change from baseline in painful score based on participants self-assessment questionnaire score (question 1) was reported. Participants were asked to rate each wound for pain/soreness in resting position as score from 0 (no pain) to 10 (severe pain).
Time Frame: Baseline, Day 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Scores on a scale
  Day 1: number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 28
  Day 1 | -0.61 (1.286) | -0.32 (0.983) | -0.46 (0.999) | -0.46 (0.922) | -0.43 (1.034) | -0.54 (1.071) | -0.39 (1.031) | -0.68 (1.219)
  Day 2: number analyzed (Participants) | 26 | 26 | 26 | 27 | 26 | 27 | 26 | 26
  Day 2 | -0.85 (1.317) | -0.42 (1.027) | -0.50 (1.140) | -0.37 (1.334) | -0.54 (1.174) | -0.44 (1.368) | -0.54 (1.140) | -0.77 (1.366)
  Day 3: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
  Day 3 | -0.93 (1.439) | -0.56 (1.188) | -0.63 (1.305) | -0.67 (1.177) | -0.67 (1.330) | -0.67 (1.387) | -0.67 (1.301) | -0.78 (1.649)
  Day 4: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
  Day 4 | -0.96 (1.400) | -0.63 (1.115) | -0.67 (1.271) | -0.70 (1.137) | -0.63 (1.391) | -0.74 (1.318) | -0.70 (1.265) | -0.81 (1.570)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change in Baseline in Painful Score with Arm Resting by Side was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p = 0.666, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.473, ANCOVA

6. Secondary Outcome: Change From Baseline in Painful Score With Arm in Normal Motion
Description: Change from baseline in Painful Score based on participants self-assessment questionnaire score (question 3) was reported. Participants were asked to rate each wound for pain/soreness in normal position as score from 0 (no pain) to 10 (severe pain).
Time Frame: Baseline, Day 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Scores on a scale
  Day 1: number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 28
  Day 1 | -0.46 (1.319) | -0.14 (0.932) | -0.29 (0.937) | -0.32 (0.863) | -0.29 (0.976) | -0.32 (0.945) | -0.32 (0.945) | -0.43 (1.069)
  Day 2: number analyzed (Participants) | 26 | 26 | 26 | 27 | 26 | 27 | 26 | 26
  Day 2 | -0.77 (1.177) | -0.35 (0.797) | -0.42 (0.857) | -0.33 (1.000) | -0.50 (0.906) | -0.33 (1.074) | -0.50 (0.860) | -0.62 (1.023)
  Day 3: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
  Day 3 | -0.74 (1.318) | -0.33 (1.000) | -0.44 (1.086) | -0.44 (1.013) | -0.52 (1.122) | -0.44 (1.121) | -0.52 (1.087) | -0.52 (1.397)
  Day 4: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
  Day 4 | -0.78 (1.251) | -0.44 (0.892) | -0.48 (1.014) | -0.52 (0.893) | -0.48 (1.156) | -0.52 (1.014) | -0.56 (1.013) | -0.56 (1.281)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline In Painful Score with Arm in Normal Motion was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p = 0.761, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.456, ANCOVA

7. Secondary Outcome: Change From Baseline in Itchy Score
Description: Change from baseline in itchy score based on participants self-assessment questionnaire score (question 5) was reported. Participants were asked to rate each wound for itchiness as score from 0 (no itch) to 10 (severe itch).
Time Frame: Baseline, Day 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Scores on a scale
  Day 1: number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 28
  Day 1 | -0.18 (1.679) | -0.21 (1.663) | -0.32 (1.588) | -0.43 (1.597) | -0.36 (1.615) | -0.25 (1.624) | -0.29 (1.630) | -0.36 (1.592)
  Day 2: number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26 | 26 | 26
  Day 2 | -0.46 (1.679) | -0.19 (1.767) | -0.31 (1.692) | -0.46 (1.679) | -0.27 (1.801) | -0.27 (1.710) | -0.27 (1.756) | -0.38 (1.675)
  Day 3: number analyzed (Participants) | 27 | 27 | 27 | 27 | 28 | 27 | 28 | 27
  Day 3 | -0.37 (1.735) | -0.19 (1.733) | -0.22 (1.717) | -0.26 (1.789) | -0.18 (2.091) | -0.04 (1.891) | -0.14 (1.840) | -0.04 (2.047)
  Day 4: number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
  Day 4 | -0.15 (1.854) | 0.00 (1.359) | -0.11 (1.826) | -0.22 (1.847) | -0.26 (1.789) | -0.11 (1.826) | -0.19 (1.841) | 0.00 (1.941)
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; Test type: Other — Change from Baseline In Itchy Score was analyzed within-treatment and between-treatment. The within-treatment comparison was performed at each post-baseline time point by comparing the post-baseline scores with the baseline score within each treatment using the paired t-test. The between-treatment comparison was performed by comparing the change from baseline between treatments using a mixed effect analysis of covariance (ANCOVA) model; p = 0.019, ANCOVA
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.325, ANCOVA

8. Primary Outcome: Time to Complete Wound Healing
Description: Time to complete wound healing: time(in days) elapsed from time of wound creation to 12 PM of day (up to Day 16) on which composite healing score(CHS) first meets complete healing criterion of being at least a score of 8 (threshold for complete healing). CHS was calculated from clinical grading of wound healing parameters as general wound appearance (0 [Poor-New or fresh wound with epithelium layer missing, wound bed appears raw and possibly oozing] to 4 [Excellent-Fully healed, skin flush against surrounding skin, slight color mismatch may be present])+smoothness (0 [Rough, uneven wound]- 4 [complete smoothness, even wound])+epithelial confluence (0 [None]- 4 [91-100%full epithelial growth]) - erythema (0 [None]- 4 [Severe]) - edema (0 [None]- 4 [Severe]) - crusting/scabbing (0 [None]- 4 [90-100% crusting/scabbing]). CHS on 25-point scale (-12 [no healing] to +12 [towards healing]) is indicative of extent of wound healing and was calculated for each wound site at each evaluation day.
Time Frame: Up to Day 16
Population: The Intent-to-Treat (ITT) set include all participants who received laser-induced wounds and started the study treatments. As planned, for this outcome measure, the data was reported for each bandage separately.
Measure: Median (Full Range); unit: Days
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Days | 11.8 [1 to 16] | 11.9 [1 to 16] | 6.9 [1 to 16] | 10.9 [1 to 16] | 5.1 [1 to 16] | 12.9 [1 to 16] | 12 [1 to 16] | 15.9 [1 to 16]
Statistical Analysis 1: Comparison: Negative Control vs Non-marketed Adhesive Bandage IP #1; All hypothesis tests was conducted at 0.05 level without adjustment of multiple comparisons; Test type: Other — Time to complete healing was analyzed using a survival analysis method. The survival function (cumulative percentage of wounds healed at each time point) was estimated by the Kaplan-Meier method for each treatment separately. The median time to complete healing was derived from the estimated survival functions and be compared using the bootstrap re-sampling method; p < 0.001, Boot-strap sampling method — no adjustments
Statistical Analysis 2: Comparison: Marketed Adhesive Bandage vs Non-marketed Adhesive Bandage IP #1; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.001, Boot-strap sampling method — no adjustments

9. Secondary Outcome: Number of Participants With Pain Duration With Arm Resting by Side
Description: Participants were asked to rate the pain as either brief, periodic, or constant in arm resting position with the Self-Assessment Questionnaire (question 2). Number of participants with pain duration (brief, periodic, or constant) with arm resting by side was reported.
Time Frame: Day 1, 2, 3 and 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Participants
  Baseline: Brief: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Brief | 18 | 21 | 20 | 21 | 20 | 19 | 19 | 19
  Baseline: Periodic: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Periodic | 2 | 0 | 3 | 2 | 1 | 2 | 2 | 3
  Baseline: Constant: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Constant | 11 | 10 | 8 | 8 | 10 | 10 | 10 | 9
  Day 1: Brief | 18 | 17 | 18 | 18 | 20 | 19 | 18 | 18
  Day 1: Periodic | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Day 1: Constant | 18 | 18 | 17 | 17 | 16 | 17 | 18 | 18
  Day 2: Brief: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Brief | 17 | 17 | 17 | 17 | 17 | 17 | 17 | 17
  Day 2: Periodic: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Periodic | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 2: Constant: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Constant | 18 | 18 | 18 | 18 | 18 | 17 | 18 | 18
  Day 3: Brief: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Brief | 16 | 16 | 16 | 16 | 16 | 15 | 16 | 15
  Day 3: Periodic: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Periodic | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Day 3: Constant: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Constant | 19 | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Day 4: Brief: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Brief | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 17
  Day 4: Periodic: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Periodic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Constant: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Constant | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 17

10. Secondary Outcome: Number of Participants With Pain Duration With Arm in Normal Motion
Description: Participants were asked to rate the pain as either brief, periodic, or constant in arm normal motion with the Self-Assessment Questionnaire (question 4). Number of participants with pain duration (brief, periodic, or constant) with arm in normal motion was reported.
Time Frame: Day 1, 2, 3 and 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Control | Marketed Adhesive Bandage | Marketed Adhesive Bandage IP-1 Benchmark Control 1 | Non-marketed Adhesive Bandage IP-Benchmark Control 2 | Non-marketed Adhesive Bandage IP #1 | Non-marketed Adhesive Bandage IP #2 | Non-marketed Adhesive Bandage IP #3 | Non-marketed Adhesive Bandage IP #4
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36
Participants
  Baseline: Brief: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Brief | 18 | 20 | 20 | 21 | 19 | 20 | 20 | 19
  Baseline: Periodic: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Periodic | 3 | 1 | 2 | 2 | 2 | 2 | 2 | 2
  Baseline: Constant: number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
  Baseline: Constant | 10 | 10 | 9 | 8 | 10 | 9 | 9 | 10
  Day 1: Brief | 17 | 17 | 18 | 18 | 19 | 19 | 18 | 18
  Day 1: Periodic | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1
  Day 1: Constant | 19 | 17 | 17 | 17 | 16 | 17 | 18 | 17
  Day 2: Brief: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Brief | 16 | 16 | 16 | 17 | 16 | 16 | 16 | 16
  Day 2: Periodic: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Periodic | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 2: Constant: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 2: Constant | 19 | 19 | 19 | 18 | 19 | 18 | 19 | 19
  Day 3: Brief: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Brief | 16 | 15 | 16 | 16 | 16 | 15 | 16 | 15
  Day 3: Periodic: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Periodic | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Day 3: Constant: number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35 | 35 | 35
  Day 3: Constant | 19 | 19 | 19 | 19 | 19 | 19 | 19 | 19
  Day 4: Brief: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Brief | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 17
  Day 4: Periodic: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Periodic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Constant: number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34 | 34 | 34
  Day 4: Constant | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 17

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety analysis population includes all participants who have IP applied at least once. As planned, adverse events were collected only on the whole participant level.
Arm/Group | All Randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 34/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized Participants (N=36)
Erythema (Skin and subcutaneous tissue disorders) | 28
Rash (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 21
Thermal burn (Injury, poisoning and procedural complications) | 2
Animal scratch (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04040933/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04040933/SAP_001.pdf